CLINICAL TRIAL: NCT06203327
Title: Atrophic Gastritis Predicts the Risk of Gastric Cancer: a Prospective Cohort Study
Brief Title: Atrophic Gastritis Predicts the Risk of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Other Study IDs: rjhy20230004
Record Dates: First submitted 2023-12-25; First posted 2024-01-12 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-12

CONDITIONS: Atrophic Gastritis
Keywords: Atrophic Gastritis; Gastric Cancer
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- OLGA 0-I
  Interventions: Other: Esophagogastroscopy (OLGA 0-Ⅰ)
- OLGA II
  Interventions: Other: Esophagogastroscopy (OLGA II)
- OLGA III-IV
  Interventions: Other: Esophagogastroscopy (OLGA III-IV)

INTERVENTIONS:
Other: Esophagogastroscopy (OLGA 0-Ⅰ) — Surveillance endoscopies at years 3-5.
  Groups: OLGA 0-I
Other: Esophagogastroscopy (OLGA II) — Surveillance endoscopies at years 2-3.
  Groups: OLGA II
Other: Esophagogastroscopy (OLGA III-IV) — Surveillance endoscopies every year.
  Groups: OLGA III-IV

SUMMARY:
Despite declining incidence rates, gastric cancer (GC) ranks the fourth leading cause of cancer-related mortality and the fifth most common cancer worldwide, with the highest incidence reported in Eastern Asia. The 5-year overall survival rate of early GC exceeds 90%, which was well above advanced GC. Most intestinal-type GCs follow the Correa cascade-inflammation,atrophy, intestinal metaplasia (IM), dysplasia and subsequent carcinoma. The presence of gastric mucosal atrophy and intestinal metaplasia are important risk factors for GC. The purpose of this study was to investigate the incidence of GC attributed to atrophic gastritis in a region with high incidence of GC.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to participate in the study and to sign and give informed consent
* Biopsies were collected based on the recommendation of updated Sydney system

Exclusion Criteria:

* under 18 or over 80 years old
* history of gastrectomy
* severe systemic diseases or malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic gastritis diagnosed by routine endoscopic screening
Sampling Method: Non-Probability Sample
Enrollment: 2042 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
early gastric neoplasm | After the baseline endoscopy, participants were scheduled for surveillance endoscopies at years 3-5 for subjects with operative link on gastritis assessment (OLGA) 0-Ⅰ, at years 2-3 for subjects with OLGA II and 1 year for subjects with OLGA III-IV.
  histological diagnosis of high-grade dysplasia, and adenocarcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No